CLINICAL TRIAL: NCT06157606
Title: Prediction Model for Inadequate Weight Loss After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: The Second Hospital of Shandong University (Other); Jining First People's Hospital (Other)
Responsible Party: Principal Investigator, Yuntao Nie, Medical doctor, China-Japan Friendship Hospital
Other Study IDs: CJBariatric001
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Bariatric Surgery; Sleeve Gastrectomy; Weight Loss
Keywords: Sleeve Gastrectomy; Weight Loss; Prediction Model
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop and validate a prediction model for estimating the probability of inadequate weight loss one year after sleeve gastrectomy.

DETAILED DESCRIPTION:
Inadequate weight loss (IWL) is a major problem after sleeve gastrectomy, leading to the recurrence of obesity-related comorbidities and increased risk of revision surgery. It is important to identify the high-risk individuals for IWL before surgery so that clinicians can initiate more rigorous weight monitoring and management strategies. Therefore, this study aims to develop a prediction model using preoperative clinical and laboratory data to estimate the risk of IWL one year after sleeve gastrectomy, and then validate it using two separate datasets.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27.5 kg/m2;
* 16 years ≤ age ≤ 70 years;
* Complete preoperative data and one-year follow-up information

Exclusion Criteria:

* Patients who did not undergo SG;
* Incomplete follow-up information;
* Patients with a history of pituitary or thyroid disease;
* Female patients who conceived within one year after surgery

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population included patients with obesity who received sleeve gastrectomy between September 2017 and September 2024. All patients were followed up for at least 1 year.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Area under receiver operating characteristic curve (AUC) of the prediction model | 1 year
  AUC reflects the discriminatory ability of the model, which was measured in this study.

SECONDARY OUTCOMES:
Brier score of the prediction model | 1 year
  Brier score reflects the calibration of the model, which was measured in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Yuntao Nie, M.D., Principal Investigator — China-Japan Friendship Hospital; Yinlu Ding, M.D., Study Director — The Second Hospital of Shandong University; Ming Zhu, M.D., Study Director — Jining First People's Hospital
Locations (1):
- Yuntao Nie, Beijing, China